CLINICAL TRIAL: NCT02223806
Title: Active Management of the Third Stage of Labour: Uterine Tonus Assessment by Midwife vs. Patient Self-administration
Acronym: UTAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Korle-Bu Teaching Hospital, Accra, Ghana (Other); University of Ghana (Other)
Responsible Party: Principal Investigator, Joyce L. Browne, Dr., UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UMC-GH 002
Record Dates: First submitted 2014-08-11; First posted 2014-08-22 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Postpartum Hemorrhage
Keywords: Postpartum hemorrhage; Uterine tonus assessment; Active management of third stage of labor
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-assessment of uterine tonus (Active Comparator): Uterine tonus assessment every 15 minutes for 2 hours by educated patient, which is standard-of-care.
  Interventions: Behavioral: Patient self-assessment of uterine tonus
- Midwife uterine tonus assessment (Experimental): Uterine tonus assessment every 15 minutes for 2 hours by midwive.
  Interventions: Behavioral: Uterine Tonus Assessment by Midwife

INTERVENTIONS:
Behavioral: Uterine Tonus Assessment by Midwife — Uterine tonus assessment every 15 minutes for 2 hours.
  Arms: Midwife uterine tonus assessment
Behavioral: Patient self-assessment of uterine tonus — Uterine tonus assessment by patient every 15 minutes for 2 hours.
  Arms: Self-assessment of uterine tonus

SUMMARY:
To determine whether there is a difference in effectiveness of routine uterine tonus assessment (every 15 minutes, for 2 hours) when performed by a midwife or self-administered by a patient on the incidence of postpartum haemorrhage, mean blood loss, and other maternal and neonatal outcomes.

DETAILED DESCRIPTION:
Rationale: Postpartum haemorrhage (PPH) is the most common cause of maternal death worldwide. The active management of the third stage of labour (AMTSL) is recognized as an effective strategy to prevent morbidity and mortality associated with PPH and reduce blood loss. AMTSL includes the provision of uterotonic drugs, controlled cord traction, delayed cord clamping and cutting, massage of the uterus, and monitoring of the uterine tonus. Although professional guidelines recommend the steps of AMTSL to be performed by health professionals, the reality of health professionals understaffed hospitals in many low- and middle income countries (LMICs) necessitates task-shifting of the final AMTSL component to patients. Yet, whether uterine tonus assessment yields the same effect when performed by patients and midwives has not been formally evaluated.

Objective: To determine whether there is a difference in effectiveness of routine uterine tonus assessment (every 15 minutes, for 2 hours) when performed by a midwife or self-administered by a patient on the incidence of postpartum haemorrhage . mean blood loss, and other maternal and neonatal outcomes.

Study design: Randomized intervention study. Study population: Pregnant women admitted in the labour to the Korle Bu Teaching Hospital, Accra, Ghana Intervention: the intervention group will receive uterine tonus assessment every 15 minutes for 2 hours by a midwife, the control group will continue the current practice of self-assessment after patient education with regular monitoring of midwives.

Main study parameters/endpoints: post-partum haemorrhage (>500 ml blood loss), severe postpartum haemorrhage (>1000 ml blood loss), mean blood loss, other maternal and neonatal outcomes.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients will receive the standard of midwifery and obstetric care, and will have access to emergency obstetric interventions. All steps of the AMTSL will be performed, with the exemption of the last step of uterine tonus assessment for which women will be randomized to receive the intervention or current practice of care. Risk associated with the intervention are discomfort because of an external assessment. Data will be obtained from record books at the ward. Women will be asked for informed consent prior to participation. This study will be approved by the Ethical en Protocol Review Committee of the University of Ghana Medical School and the Medical Ethical Research Committee of the University Medical Center Utrecht.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Be in labor with an expected vaginal delivery, as assessed by the midwives
* Gestation age ≥ 37 weeks
* Received antenatal instructions on postnatal uterine tonus assessment
* Provided informed consent.

Exclusion Criteria:

* Age <18
* Elective caesarean delivery
* Severe anemia (<8g/dL)
* Placenta praevia
* Anticipated breech delivery
* Referred patients who have not received antenatal care (ANC) uterine tonus assessment instructions
* Multiple Pregnancy
* Intra uterine fetal death

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 800 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Postpartum hemorrhage (>500 ml blood loss) | within 24 hours postpartum
  To determine whether there is a difference in effectiveness of routine uterine tonus assessment (every 15 minutes, for 2 hours) to prevent post-partum hemorrhage (≥500 ml blood loss) when performed by a midwife and self-administered by a patient.

SECONDARY OUTCOMES:
Mean blood loss (in ml) | Within 24 hours postpartum
Severe post-partum hemorrhage | Within 24 hours postpartum
  >1000ml blood loss
Use of additional uterotonics | Within 24 hours postpartum
Use of other procedures for management of postpartum hemorrhage | Within 24 hours postpartum
  I.e. surgery, manual placenta tissue removal
Late postpartum hemorrhage | From 24 hours and upto one week
  Based on readmission

CONTACTS AND LOCATIONS:
Overall Officials: Joyce L Browne, MD, MSc, Principal Investigator — UMC Utrecht, the Netherlands; Kerstin D Klipstein-Grobusch, PhD MSc, Principal Investigator — University Medical Center Utrecht, The Netherlands; Nelson Damale, MBChB, Principal Investigator — Korle-Bu Teaching Hospital, Accra, Ghana
Locations (1):
- Korle Bu Teaching Hospital, Accra, Ghana

REFERENCES:
- [Derived] Browne JL, Damale NK, Raams TM, Van der Linden EL, Maya ET, Doe R, Rijken MJ, Adanu R, Grobbee DE, Franx A, Klipstein-Grobusch K. Uterine Tonus Assessment by Midwives versus Patient self-assessment in the active management of the third stage of labor (UTAMP): study protocol for a randomized controlled trial. Trials. 2015 Dec 18;16:580. doi: 10.1186/s13063-015-1111-5. PMID 26683621